CLINICAL TRIAL: NCT00230763
Title: Determination Of Predictive Factors Allowing To An Additional 10% Reduction Of Intra-Ocular Pressure After A 12-Week Treatment With Latanoprost 0.005% / Timolol 0.5% Fixed Combination (Xalacom) In Previously Treated Patients With Open Angle Glaucoma Or Ocular Hypertension
Brief Title: Determination Of Predictive Factors Allowing To An Additional 10% Reduction Of Intra-Ocular Pressure
Acronym: PREDICOM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6641040
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2015-03

CONDITIONS: Glaucoma, Primary Open Angle (POAG); Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost; Timolol; Xalacom; Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: LATANOPROST 0.005% / TIMOLOL 0.5% FIXED COMBINATION
- Procedure (Other)
  Interventions: Procedure: GSS questionnaire; Procedure: IOP; Procedure: Visual acuity

INTERVENTIONS:
Procedure: GSS questionnaire — D0, D30 and D84
  Arms: Procedure
Procedure: IOP — D0, D30 and D84
  Arms: Procedure
Drug: LATANOPROST 0.005% / TIMOLOL 0.5% FIXED COMBINATION — in the evening during 84 days
  Other Names: XALACOM
  Arms: Active
Procedure: Visual acuity — D0 and D84
  Arms: Procedure

SUMMARY:
To determine the predictive factors of a positive response to latanoprost 0.005% / timolol 0.5% fixed combination (defined as a 10% IOP reduction from baseline), after 12 weeks of treatment (age, sex, ethnic origin, patient's medical history, family history of OAG or OHT, concomitant systemic treatment with beta-blockers, etiology, IOP at baseline, corneal thickness, compliance, and adverse events).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients,
* Aged > than equal to 18 years,
* Patient presenting with an OHT or OAG with an IOP � 21 mmHg,
* Patient currently treated with ophthalmic beta-blockers monotherapy and requiring a change of the ophthalmic medication due to insufficient response to treatment,

Exclusion Criteria:

* Patient currently treated by or having received within the last month any ophthalmic hypotensive agent other than a beta-blocker,
* Patient presenting any contraindication to latanoprost or timolol,
* Patient with history of asthma, obstructive broncho-pneumopathy, sinusal bradycardia (pulse rate < 60 bpm), auriculo-ventricular block, cardiac insufficiency, Raynaud disease or any other condition that would preclude the patient from taking the prescribed medication,
* Patient with known intolerance to benzalkonium chloride or any excipient contained in the trial treatment,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2005-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
A positive response defined as an additional IOP reduction over 10% after 12 weeks of treatment in the intent to treat (ITT) population. | after 12 weeks of treatment

SECONDARY OUTCOMES:
Absolute and relative IOP change after 4 and 12 weeks of treatment | week 4 and 12
Percentage of patients achieving a target IOP value: under 18 mmHg and under 16 mmHg after 12 weeks of treatment, | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (93):
- France (93):
  - Pfizer Investigational Site, Agen
  - Pfizer Investigational Site, Amboise
  - Pfizer Investigational Site, Amiens
  - Pfizer Investigational Site, Andrésy
  - Pfizer Investigational Site, Asnières-sur-Seine
  - Pfizer Investigational Site, Aubière
  - Pfizer Investigational Site, Aurillac
  - Pfizer Investigational Site, Belfort
  - Pfizer Investigational Site, Besançon
  - Pfizer Investigational Site, Béziers
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Bourg-en-Bresse
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Cannes
  - Pfizer Investigational Site, Castelsarrasin
  - Pfizer Investigational Site, Chalon-sur-Saône
  - Pfizer Investigational Site, Chamalieres-Royat
  - Pfizer Investigational Site, Chambéry
  - Pfizer Investigational Site, Chartres
  - Pfizer Investigational Site, Chassieu
  - Pfizer Investigational Site, Châlons-en-Champagne
  - Pfizer Investigational Site, Château-Renault
  - Pfizer Investigational Site, Châteaudun
  - Pfizer Investigational Site, Clamart
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Colmar
  - Pfizer Investigational Site, Coulommiers
  - Pfizer Investigational Site, Dax
  - Pfizer Investigational Site, Étampes
  - Pfizer Investigational Site, Figeac
  - Pfizer Investigational Site, Fréjus
  - Pfizer Investigational Site, Goussainville
  - Pfizer Investigational Site, Haguenau
  - Pfizer Investigational Site, Hyères
  - Pfizer Investigational Site, Issy-les-Moulineaux
  - Pfizer Investigational Site, Ivry-sur-Seine
  - Pfizer Investigational Site, Jarny
  - Pfizer Investigational Site, La Flèche
  - Pfizer Investigational Site, Langon
  - Pfizer Investigational Site, Lannion
  - Pfizer Investigational Site, Le Mans
  - Pfizer Investigational Site, Le Quesnoy
  - Pfizer Investigational Site, Les Clayes-sous-Bois
  - Pfizer Investigational Site, Les Lilas
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Limoges
  - Pfizer Investigational Site, Luxeuil-les-Bains
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Meaux
  - Pfizer Investigational Site, Meudon
  - Pfizer Investigational Site, Meyzieu
  - Pfizer Investigational Site, Montargis
  - Pfizer Investigational Site, Montbéliard
  - Pfizer Investigational Site, Montigny-le-Bretonneux
  - Pfizer Investigational Site, Moulins
  - Pfizer Investigational Site, Mulhouse
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Nemours
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Nœux-les-Mines
  - Pfizer Investigational Site, Orléans
  - Pfizer Investigational Site, Orsay
  - Pfizer Investigational Site, Pantin
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Pau
  - Pfizer Investigational Site, Perpignan
  - Pfizer Investigational Site, Poissy
  - Pfizer Investigational Site, Quetigny
  - Pfizer Investigational Site, Rillieux-la-Pape
  - Pfizer Investigational Site, Roanne
  - Pfizer Investigational Site, Roquebrune-Cap-Martin
  - Pfizer Investigational Site, Roye
  - Pfizer Investigational Site, Saint-Girons
  - Pfizer Investigational Site, Saint-Laurent-du-Var
  - Pfizer Investigational Site, Saint-Maur-des-Fossés
  - Pfizer Investigational Site, Saint-Quentin
  - Pfizer Investigational Site, Sainte-Maure-de-Touraine
  - Pfizer Investigational Site, Saintes
  - Pfizer Investigational Site, Salon-de-Provence
  - Pfizer Investigational Site, Sceaux
  - Pfizer Investigational Site, Toulon
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Tremblay-en-France
  - Pfizer Investigational Site, Troyes
  - Pfizer Investigational Site, Vauvert
  - Pfizer Investigational Site, Vendôme
  - Pfizer Investigational Site, Versailles
  - Pfizer Investigational Site, Viarmes
  - Pfizer Investigational Site, Villeneuve-la-Garenne
  - Pfizer Investigational Site, Villeparisis
  - Pfizer Investigational Site, Villiers-le-Bel
  - Pfizer Investigational Site, Wasselonne

REFERENCES:
- [Derived] Sellem E, Rouland JF, Baudouin C, Bron A, Denis P, Nordmann JP, Renard JP. Predictors of additional intraocular pressure reduction in patients changed to latanoprost/timolol fixed combination. BMC Ophthalmol. 2010 Mar 26;10:10. doi: 10.1186/1471-2415-10-10. PMID 20346127
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6641040&StudyName=Determination%20Of%20Predictive%20Factors%20Allowing%20To%20An%20Additional%2010%25%20Reduction%20Of%20Intra-Ocular%20Pressure